CLINICAL TRIAL: NCT06694662
Title: PKU EASY Microtabs Plus - Acceptability and Tolerance
Acronym: PEMP-AT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galen Limited (Industry)
Collaborators: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-004
Record Dates: First submitted 2024-11-12; First posted 2024-11-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Phenylketonuria (PKU)
Keywords: PKU; Microtabs; protein substitute; amino acid
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): All participants will be assessed by their dietitian and prescribed an appropriate amount of the study product, PKU EASY Microtabs Plus, to manage their phenylketonuria.
  Interventions: Dietary Supplement: PKU EASY Microtabs Plus

INTERVENTIONS:
Dietary Supplement: PKU EASY Microtabs Plus — PKU EASY Microtabs Plus is a food for special medical purposes (FSMP). This product is for use in the dietary management of Phenylketonuria (PKU) in patients from 3 years of age upwards.
  PKU EASY Microtabs Plus is a microtablet form, slow-release, phenylalanine-free protein substitute containing a blend of essential and non-essential amino acids, vitamins, minerals and trace elements.

SUMMARY:
PEMP-AT is a prospective, single-arm, open-label, 1-week acceptability study to evaluate PKU EASY Microtabs Plus for the dietary management of participants with phenylketonuria (PKU). Up to 10 participants aged 3 years and above will be recruited in a single-centre in the UK.

DETAILED DESCRIPTION:
PKU is a rare inborn error of metabolism with a prevalence of 1 in 10,000 in the UK population. The mainstay of treatment for most individuals is dietary therapy with a strict protein-restricted diet. We propose to recruit children with a diagnosis of PKU aged 3 years and above.

The study product, PKU EASY Microtabs Plus is a food for special medical purposes (FSMP), as defined by the Delegated Act EU 2016/128, used for the dietary management of Phenylketonuria (PKU).

The study will be investigating the acceptability of PKU EASY Microtabs Plus, as defined by the Advisory Committee on Borderline Substances (ACBS). This includes the following:

participant adherence to recommended intakes gastrointestinal symptoms evaluations of palatability. Each participant will be on the study for 1 week.

The study consists of a 1 week period where participants introduce the study product into their diet. Gastrointestinal tolerance, compliance and product acceptability will be evaluated.

Data collection will be performed using paper data collection forms completed by the investigators at the baseline and end of study visits. Patients/parents/guardians, as appropriate, will also complete a brief daily questionnaire on each of the 7 study days. There will also be a questionnaire completed by the patient/parents/guardians over the course of the study, in relation to protein substitute intake, gastrointestinal tolerance, and product acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU requiring an appropriate protein substitute
* Subjects who are already taking an appropriate protein substitute and are willing to try the study product for 7 days
* Subjects aged 3 years and above
* Written informed consent obtained from subject or parent/legal guardian, depending on subject age

Exclusion Criteria:

* Presence of serious concurrent illness
* Lead Dietitian's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study, with the exception of sapropterin
* Any subject having taken antibiotics over the previous 2 weeks leading up to the study
* Subjects less than 3 years of age

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Change in GI tolerance (participant) | Week 0, week 1
  Gastrointestinal tolerance assessed using symptom and severity questionnaire completed by the participants. Severity of symptoms will be rated on a scale of 0 - 3, with 0 being no symptoms and 3 being severe or very troublesome symptoms.
Rate of patient compliance with consumption of the prescribed volume of study product | Week 1
  Assessed via participant diary regarding study product intake. The quantity of study product actually consumed vs the prescribed amount will be recorded. The reason for not consuming the full dose will be recorded by the patient/parent/guardian as free text.
Change in product acceptability | Week 1
  Assessed via a product acceptability questionnaire completed by the participant/parent/guardian. Organoleptic properties, such as taste and texture, of the study product will be assessed on a rating scale of terrible to great.

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Ph.D., Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (1):
- Birmingham Children's Hospital, Birmingham, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the very small number of participants and rarity of the condition being tested the ability to maintain participant pseudonymity could be compromised.